CLINICAL TRIAL: NCT03490994
Title: Rivaroxaban Once Daily Versus Dose-adjusted Vitamin K Antagonist on the Biomarkers in Acute Decompensated Heart Failure and Atrial Fibrillation (ROAD HF-AF)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0776
Record Dates: First submitted 2018-03-11; First posted 2018-04-06 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — Rivaroxaban; Warfarin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: warfarin vs. rivaroxaban
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental): Rivaroxaban
  Interventions: Drug: Rivaroxaban
- Warfarin (Active Comparator): warfarin + enoxaparin
  Interventions: Drug: Warfarin + LMWH

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 20mg qd (15mg qd when CrCl 30-49 ml/min using creatinine-based CKD-EPI equations) for 6 months
  Arms: Rivaroxaban
Drug: Warfarin + LMWH — dose-adjusted warfarin (target INR 2-3) for 6 months + LMWH (enoxaparin 1 mg/kg q12h for a few days until INR target achieved) if indicated
  Arms: Warfarin

SUMMARY:
Vitamin K antagonists (VKAs) are used to reduce the risk of stroke (cerebral vascular dysfunction) in AF patients. However, VKAs interact with drugs/food and the drug level is influenced by worsening of renal function, liver congestion or hemodynamic alterations in acute decompensated heart failure (ADHF). New oral anticoagulants (rivaroxaban, apixaban, dabigatran) are alternatives to VKA, such as warfarin. In post hoc analysis of ROCKET AF trial, 63.7% patients had HF and treatment-related outcomes were similar in patients with and without HF (Circulation HF. 2013; 6:740-7). So rivaroxaban 20 mg daily (or 15 mg daily in patients with creatinine clearance 30-49 mL/min) was safe in nonvalvular AF patients with HF. However, the clinical effect and safety of rivaroxaban were largely unknown in acute decompensated heart failure (ADHF) patients with atrial fibrillation (AF).

ROAD HF-AF is the exploratory study to assess the change of surrogate markers (hsTn, d-dimer) when treated with rivaroxaban vs. warfarin and to strengthen the basis for future biomarker-based therapy in ADHF patients

ELIGIBILITY:
Inclusion Criteria:Hospitalized patients with a primary diagnosis of ADHF with AF One of the following criteria and LVEF ≤ 40% (at least 1 year before admission or admission)

1. dyspnea at rest
2. tachypnea; a respiratory rate > 20/min
3. rales
4. pulmonary edema on chest X-ray

Exclusion Criteria:

1. History of increased bleeding risk (like ROCKET AF exclusion criteria)
2. Contraindication to anti-coagulation therapy
3. ACS diagnosis
4. Hospitalization plan for PCI, coronary artery bypass graft surgery, other cardiac invasive interventions (e.g. catheter ablation, pacemaker, CRT, ICD implantation)
5. Currently on dual anti-platelet therapy (aspirin + ADP receptor antagonist) or single antiplatelet therapy with a novel AP (e.g. Ticagrelor, Prasugrel)
6. Cardiogenic shock (systolic blood pressure, SBP, < 80 mmHg)
7. Patients with CrCl < 30 ml/min using creatinine-based CKD-EPI equations
8. Elevated liver enzymes (3 times over upper reference limit) or liver cirrhosis
9. Uncontrolled hypertension (SBP > 180 mmHg)
10. Allergy, adverse drug reaction, hypersensitivity to rivaroxaban or warfarin
11. Life expectancy < 6 months (e.g. metastatic malignancy)
12. Pregnancy, or women of childbearing age

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
the change of high sensitive troponin | Baseline to 72 hours
  The maximum hsTn value change from baseline to during hospitalization

SECONDARY OUTCOMES:
1) the change of hish sensitive troponin | 1) On admission, hospital day #2, hospital day #4, hospital day #7 or discharge, 1 month/6month after discharge
  1) The change from baseline in hsTn on Day2, day4, day7 (or discharge), and follow-up visits at 1 month, 6 months
2) the change of D-dimer | 2) On admission, hospital day #2, hospital day #4, hospital day #7 or discharge, 1 month/6month after discharge
  2) D-dimer change from baseline during hospitalization (day2, day4, day7 or discharge) & follow-up visits at 1, 6 months
3) the change of NT-proBNP | 3) On admission, hospital day #7 or discharge, 1 month/6month after discharge
  3) TAT complex, PAI-1, hsCRP, NT-proBNP, sST2, galectin-3, cystatin C, NGAL, NAG change from baseline to day7 or discharge & 1,6 months after discharge
4) bleeding event | 4) On admission, hospital day #2, hospital day #4, hospital day #7 or discharge, 1 month/3month/6month after discharge
  4) Incidence proportion and rate of major/minor bleeding during the study
5) hospital stay | 5) The duration of hospital stay, average 7 days
  5) Length of hospital stay
6) all-cause mortality | 6) 6 months after hospitalization
  6) Incidence proportion of in-hospital all-cause death cases
7) all-cause hospitalization & mortality | 7) 6 months after hospitalization
  7) Time to the first composite event of all-cause mortality or cardiovascular re-hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No